CLINICAL TRIAL: NCT04415099
Title: The Effect of Tibialis Posterior Muscle Fatigue on Plantar Pressure Characteristics
Brief Title: Tibialis Posterior Fatigue and Plantar Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pınar Kısacık, PhD, Research Assistant, PhD., Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: LUT 12/46-16
Record Dates: First submitted 2020-04-14; First posted 2020-06-04 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-05

CONDITIONS: Muscle Fatigue
Keywords: Plantar pressure distribution; muscle fatigue; tibialis posterior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One group (Experimental): Only one group was assessed before and after performing muscle fatigue protocol.
  Interventions: Other: Muscle fatigue protocol

INTERVENTIONS:
Other: Muscle fatigue protocol — Tibialis posterior was fatigued using 2 exercises:
  1. Unilateral heel raise exercise
  2. Close chain resisted foot adduction exercise

SUMMARY:
The purpose of this study is to find out the changes in the measurable parameters of the dynamic and static position of the foot, caused by the tibialis posterior muscle which is activated by the fatigue protocol. The study includes 30 healthy patients whose socio-demographic and descriptive characteristics are held. The changes in the dynamic and static position of foot were measured by pedobarography whereas the level of fatigue was measured by Borg Fatigue Scale.

DETAILED DESCRIPTION:
The purpose of this study is to find out the changes in the measurable parameters of the dynamic and static position of the foot, caused by the tibialis posterior muscle which is activated by the fatigue protocol. The study includes 30 healthy patients whose socio-demographic and descriptive characteristics are held. The changes in the dynamic and static position of foot were measured by pedobarography whereas the level of fatigue was measured by Borg Fatigue Scale. The variables were investigated using Shapiro-Wilk's test to determine the normality. The student's t-test for paired samples were used to analyse, means (X), standard deviations (SD), 95% confidence intervals (95%CI), mean difference and Cohen's d-effect size were calculated. The significance level was set at .05. The effect size was considered 'small' if d= .20; 'medium' if .d=.5; 'large' if d= .8.

ELIGIBILITY:
Inclusion Criteria:

* All participants were currently free from congenital or traumatic deformity to either lower extremity,
* A history of foot pain,
* Prior history of surgery to the foot and lower extremity
* A traumatic injury to the ankle or foot 12 months prior to the start of data collection.

Exclusion Criteria:

* Participants were excluded from this study if they had any orthopedic or neurological disorder, need to use an assistive device or orthoses.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Peak Plantar Pressures of the foot | 1 month
  The plantar pressure profiles were divided into 10 anatomical regions by using software support. These regions corresponded to followings : hallux (toe1), toes 2-5, first to fifth metatarsals (Meta1, Meta2, Meta3, Meta4, and Meta5), mid foot (MF), medial heel (MH), and lateral heel (LH). Peak pressure (PP, Newton-N) was analysed for all regions separately.

SECONDARY OUTCOMES:
Contact area of the foot | 1 month
  The percentage of the contact area (CA%) of forefoot (FF), midfoot (MF) and hindfoot (HF) was recorded. The right foot of each subjects was chosen to be analysed to maintain independence of data. In line with this, all tests' first and third trials were exculeded from statistical analysis, because of avoiding acclimatization and boredom or tiredness.
Foot axis angle | 1 month
  Foot axis angle (FAA) was recorded in unit of degree (o). The right foot of each subjects was chosen to be analysed to maintain independence of data. In line with this, all tests' first and third trials were exculeded from statistical analysis, because of avoiding acclimatization and boredom or tiredness.
Subtalar angle | 1 month
  Minimum and maximum value of the subtalar angle (STA) was recorded in unit of degree (o). The right foot of each subjects was chosen to be analysed to maintain independence of data. In line with this, all tests' first and third trials were exculeded from statistical analysis, because of avoiding acclimatization and boredom or tiredness.
Static plantar pressure | 1 month
  The plantar pressure profiles were divided into 10 anatomical regions by using software support. These regions corresponded to followings : hallux (toe1), toes 2-5, first to fifth metatarsals (Meta1, Meta2, Meta3, Meta4, and Meta5), mid foot (MF), medial heel (MH), and lateral heel (LH). Peak pressure (PP, Newton-N) was analysed for all regions separately.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Bek, Prof.Dr., Study Director — Lokman Hekim University; Azize Reda Caferoglu Tunç, MSc, Principal Investigator — Lokman Hekim University
Locations (1):
- Pınar Kısacık, Ankara, Turkey (Türkiye)